CLINICAL TRIAL: NCT01678651
Title: Embryo Kinetcis From Embryos Deriving From Egg Donation Cycle With Different Stimulation Protocol: Recombinant FSH vs Human FSH
Brief Title: Embryo Kinetics and Stimulation Protocol: Recombinant Follicle Stimulating Hormone (FSH) Versus Human FSH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: IVI Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAD-NB-08-2012-01
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2015-03

CONDITIONS: Embryo Kinetics
Keywords: time-lapse, FSH, kinetics
MeSH Terms: interventions — Follicle Stimulating Hormone, Human

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Human FSH (Active Comparator): Human FSH
  Interventions: Procedure: Stimulation with human FSH
- Recombinant FSH (Active Comparator): Recombinant FSH
  Interventions: Procedure: Stimulation with recombinant FSH

INTERVENTIONS:
Procedure: Stimulation with human FSH — Human FSH
  Arms: Human FSH
Procedure: Stimulation with recombinant FSH — Recombinant FSH
  Arms: Recombinant FSH

SUMMARY:
Different kinetics markers have been proposed to select embryos with higher implantation rates. The effect of external factors on these markers, such as the stimulation protocol should be analyzed. There are two different types of FSH that are commonly used for in vitro fertilization (IVF) in egg donation cycles, recombinant FSH and human FSH. The effect of each kind of hormone on embryo kinetcis is still unknown. The aim of this study is to observe if there is a difference in embryo kinetics and morphology as well as oocyte morphological parameters between the two types of FSH and therefore to analyze if such markers can be used despite of the stimulation protocols chosen.

ELIGIBILITY:
Inclusion Criteria:

•Egg donation cycles with more than 8MII in oocyte retrieval day

Exclusion Criteria:

* Male factor
* Uterine malformations
* genetic alterations

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
time of cell cleavage | February 2012
  Analysis of cell cleavage

SECONDARY OUTCOMES:
Embryo and oocyte morphology | February 2012
  Analysis of all oocytes
Outcome rates (implantation, pregnancy and miscarriage rate) | February 2012
  Time requierd to know all the implantation, pregnancy and miscarriage rate

CONTACTS AND LOCATIONS:
Locations (1):
- Insituto Valenciano de Infertilida, Madrid, Madrid, Spain